CLINICAL TRIAL: NCT01886430
Title: Effects of Low-frequency Electrical Stimulation in Sympathetic Nerve Activity and Peripheral Vasoconstriction in Patients With Advanced HF
Brief Title: Effects of Low-frequency Electrical Stimulation in Patients With Advanced HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Raphaela Vilar Ramalho Groehs, PhD student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FES
Record Dates: First submitted 2013-04-09; First posted 2013-06-25 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Electrical Stimulation (Experimental): Functional Electrical Stimulation for 10 days
  Interventions: Other: Functional electrical stimulation
- Control Electrical Stimulation (Placebo Comparator): Control Electrical Stimulation for 10 days
  Interventions: Other: Placebo electrical stimulation

INTERVENTIONS:
Other: Functional electrical stimulation — Functional electrical stimulation for 10 days
  Arms: Functional Electrical Stimulation
Other: Placebo electrical stimulation — Placebo electrical stimulation for 10 days
  Arms: Control Electrical Stimulation

SUMMARY:
The purpose of this study is to verify the effects of low frequency functional electrical stimulation in heart failure patients hospitalized for treatment of the syndrome.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of low frequency functional electrical stimulation on control autonomic and peripheral function in heart failure patients hospitalized for treatment of the syndrome. A randomized clinical trial with 30 advanced heart failure patients will be randomly assigned to functional electrical stimulation (Functional EE, n= 15) e 2) sensory electrical stimulation (Sensory EE, n=15). The functional electrical stimulation will be applied in the rectus femoris, and gastrocnemius, with frequency of 10 Hz, pulse duration of 150 ms, stimulation time (time on) of 20 seconds, resting time (time off) of 20 seconds and intensity according to the discomfort threshold of the patient , checked every day until achieve a maximum of 70mA. The session will last 60 minuts. It will be held every weekday for a period of 10 days. The effects of interventions on functional capacity, autonomic control, peripheral function, peripheral muscle strength and quality of life will be analyzed at baseline and at the end of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced heart failure,
* Class Functional IV, according to the criteria of New York Heart Association (NYHA),
* Aged over 18 years,
* Etiology hypertensive, ischemic, idiopathic or chagas disease,
* Left ventricular ejection fraction ≤ 30%.

Exclusion Criteria:

* Patients with hypertension lung disease and oxygen-dependent,
* Neurological and neuromuscular disease that presenting paresthesia or plegia of the lower limbs,
* Insulin-dependent diabetes mellitus (type I),
* Peripheral arterial occlusive disease,
* Peripheral neuropathy,
* Use of pacemaker or implantable cardiodefibrillator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional assessment | 10 days
  To assess the effects of the functional electrical stimulation in patients with advanced heart failure.

SECONDARY OUTCOMES:
Peripheral function | 10 days
  To assess the effects of the functional electrical stimulation in patients with advanced heart failure.
Peripheral muscle strength | 10 days
  To assess the effects of the functional electrical stimulation in patients with advanced heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - HC/FMUSP, São Paulo, São Paulo, Brazil